CLINICAL TRIAL: NCT04009681
Title: An Open-Label, Multicenter Phase 1/2 Dose Escalation and Expansion Study of THOR-707 as a Single Agent and as a Combination Therapy in Adult Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Study Evaluating Safety and Therapeutic Activity of THOR-707 in Adult Subjects With Advanced or Metastatic Solid Tumors (THOR-707-101)
Acronym: HAMMER
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated as per Sponsor decision. The decision was not related to any safety concerns.
Sponsor: Synthorx, Inc, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: THOR-707-101 (TCD16843); U1111-1298-7281 (Other: WHO ICTRP); 2023-508422-95-00 (Other: EMA)
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Metastasis
Keywords: Synthorx; THOR-707; THOR 707; Interleukin 2; Interleukin-2; IL2; oncology; immuno-oncology; immunotherapy; IL-2; SAR444245; Sanofi
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — pembrolizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort A-THOR-707 Q2W Monotherapy (Dose Escalation) (Experimental): Subjects with advanced or metastatic solid tumors will receive THOR-707 in sequential ascending doses as a monotherapy via intravenous (IV) administration every 2 weeks (Q2W) until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: THOR-707
- Cohort B-THOR-707 Q3W Monotherapy (Dose Escalation) (Experimental): Subjects with advanced or metastatic solid tumors will receive THOR-707 in sequential ascending doses as a monotherapy via IV administration every 3 weeks (Q3W) until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: THOR-707
- Cohort C-THOR-707 Q3W with checkpoint inhibitor (Dose Escalation) (Experimental): Subjects with advanced or metastatic solid tumors will receive THOR-707 Q3W in sequential ascending doses in combination with a checkpoint inhibitor Q3W or every 6 weeks (Q6W) via IV administration until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: THOR-707; Drug: Checkpoint inhibitor
- Cohort D-THOR-707 Q3W with anti-EGFR antibody (Dose Escalation) (Experimental): Subjects with advanced or metastatic solid tumors will receive THOR-707 Q3W in sequential ascending doses in combination with an anti-EGFR antibody weekly dosing (QW) via IV administration until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: THOR-707; Drug: anti-EGFR antibody
- Cohort E-THOR-707 Q2W with checkpoint inhibitor (Dose Expansion) (Experimental): Subjects with advanced or metastatic solid tumors will receiveTHOR-707 Q2W at recommended Phase 2 dose (RP2D) with a checkpoint inhibitor via IV administration Q6W; it will consist of one 8-week cycle of THOR-707 monotherapy on Cycle 1 Day 1 followed by THOR-707 Q2W + checkpoint inhibitor Q6W starting at Cycle 1 Day 15. Subsequently treatment will consist of repeated 6-week cycles with combination therapy.
  Interventions: Drug: THOR-707; Drug: Checkpoint inhibitor
- Cohort F-THOR-707 Q3W with checkpoint inhibitor (Dose Expansion) (Experimental): Subjects with advanced or metastatic solid tumors will receive THOR-707 Q3W at recommended Phase 2 dose (RP2D) with a checkpoint inhibitor via IV administration Q6W will consist of one 9-week cycle of THOR monotherapy on Cycle 1 Day 1 followed by THOR-707 Q3W + checkpoint inhibitor at Cycle 1 Day 22. Subsequently treatment will consist of repeated 6-weeks cycles with combination therapy.
  Interventions: Drug: THOR-707; Drug: Checkpoint inhibitor
- Cohort G Monotherapy QW/Q2W (Dose Escalation) (Experimental): Subjects with advanced or metastatic solid tumors will receive THOR707 monotherapy QW for 6 weeks (induction period), and then every Q2W (maintenance period), which is referred as QW/Q2W thereafter, until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: THOR-707
- Cohort H Monotherapy QW/Q2W (Dose Expansion) (Experimental): Subjects with late-line metastatic melanoma will receive THOR707 monotherapy at RP2D for Cohort G. Cycle 1 will consist of THOR-707 QW for 6 weeks; Cycle 2 and beyond will consist of THOR-707 Q2W.
  Interventions: Drug: THOR-707

INTERVENTIONS:
Drug: THOR-707 — Pharmaceutical form: solution for intravenous (IV) administration; Route of administration: IV administration
  Other Names: SAR444245; Pegenzileukin
Drug: Checkpoint inhibitor — Pharmaceutical form: solution for IV administration; Route of administration: IV administration
  Other Names: pembrolizumab
  Arms: Cohort C-THOR-707 Q3W with checkpoint inhibitor (Dose Escalation); Cohort E-THOR-707 Q2W with checkpoint inhibitor (Dose Expansion); Cohort F-THOR-707 Q3W with checkpoint inhibitor (Dose Expansion)
Drug: anti-EGFR antibody — Pharmaceutical form: solution for IV administration; Route of administration: IV administration
  Other Names: cetuximab
  Arms: Cohort D-THOR-707 Q3W with anti-EGFR antibody (Dose Escalation)

SUMMARY:
Primary Objectives:

* Evaluate the safety and tolerability of THOR-707 as a single agent and as a combination therapy (identify Dose Limiting Toxcitiy (DLTs) in Cohorts A, B, C, D, and G, and adverse events (AEs)/serious adverse event (SAE) profile in Cohorts A, B, C, D, E, F, and G)
* Define the Maximium Tolerated Dose (MTD) and/or the Recommended Phase 2 Dose (RP2D) of THOR-707 as a single agent and as a combination therapy (Cohorts A, B, C, D, and G)
* Evaluate preliminary anti-tumor activity of THOR-707 as a single agent by determination of the objective response rate (ORR) defined according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (Cohort H only)

Secondary Objectives:

* Evaluate preliminary anti-tumor activity of THOR-707 as a single agent and as a combination therapy by determination of the objective response rate (ORR) defined according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (Cohorts A, B, C, D, E, F, and G)
* Determine time to response (TTR), duration of response (DOR), progression-free survival (PFS), overall survival (OS), disease control rate (DCR), and clinical benefit rate (CBR) of THOR-707 as a single agent and as a combination therapy
* Evaluate the safety and tolerability of THOR-707 monotherapy QW/Q2W (AE/serious adverse event [SAE] profile) (Cohort H only).

DETAILED DESCRIPTION:
The study duration per participant is approximately 24 months (inclusive of follow-up). Cohorts A, B, C, and D have been completed.

ELIGIBILITY:
Key Inclusion Criteria:

* Measurable disease per RECIST v1.1. For Cohort G participants must have at least 1 measurable lesion, and for Part 3 (Cohorts E, F and H) participants must have at least 2 measurable lesions to safely perform mandatory pre & on-treatment biopsy.
* Life expectancy greater than or equal to 12 weeks.
* For Part 2 exclusively: While it is highly preferred to enroll subjects who are naïve to PD-1 inhibitors into a Part 2 dose escalation cohort, this is not an enrollment requirement. However, subjects who enroll into a Part 2 safety expansion cohort must be naïve to PD-1 inhibitors. If such subject is unable to meet this requirement but otherwise remains a good candidate for study enrollment, the Investigator should discuss with the Sponsor whether the subject may be enrolled.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate cardiovascular, hematological, liver, and renal function.
* Histologically or cytologically confirmed diagnosis of advanced and/or metastatic solid tumors with at least one tumor lesion with location accessible to safely biopsy per clinical judgment of the Investigator.

  * Caution: Cohort D only patients with KRAS mutant colon cancer have not typically benefitted from the addition of cetuximab in earlier lines of therapy.
  * Caution: Cohorts E & F enrollment will include only patients with tumors for which anti-PD(L)1 as single agent or in combination treatments are approved.
  * Caution: For Cohort H, the participant must have received at least one prior line of therapy for metastatic melanoma and/or does not have any standard of care (SoC) treatment option or participant declines or is intolerant to be treated with SoC treatment.
* Subjects with advanced or metastatic solid tumors who have refused SoC; or for whom no reasonable SoC exists that would confer clinical benefit; or for whom standard therapy is intolerable, not effective, or not accessible.
* Prior anti-cancer therapy is allowed as long as any treatment related toxicity is resolved to an appropriate level.
* Females of childbearing potential and men who are not surgically sterile must agree to use medically-accepted method of birth control during the study and for at least7 days (for Cohorts A, B, G and H), at least 2 months (for Cohort D), or at least 4 months (for Cohorts C, E and F) for females, and for at least 3 days for males [corresponding to the time needed to eliminate study intervention] after the last dose of study intervention.
* [Females] Negative serum pregnancy test within 7 days prior to initiating study treatment in premenopausal women and women less than 12 months after menopause.
* [Males] Agreement to refrain from donating or banking sperm during the treatment period and for at least 3 days after last dose of study treatment.
* In Spain, Chile, and Argentina: Only cohorts G and H will be open to enrollment.

Key Exclusion Criteria:

* Radiotherapy ≤ 14 days prior to first dose of study drug (palliative radiation or stereotactic radiosurgery within 7 days prior to start of study treatment).
* Treated with systemic anti-cancer therapy or an investigational agent within 2 weeks prior to start of study drug treatment (within 4 weeks for immunotherapy and tyrosine kinase inhibitor therapy).
* Subjects who experienced Grade 3 or higher immune-related toxicity from prior immuno-oncology therapy.
* Major surgery ≤ 30 days prior to first dose of study drug, or has not recovered to at least Grade 1 from adverse effects from such procedure, or anticipation of the need for major surgery during study treatment.
* Active autoimmune disease requiring systemic treatment within the past 3 months or have a documented history of clinically severe autoimmune disease that requires systemic steroids or immunosuppressive agents.
* Primary central nervous system (CNS) disease or leptomeningeal disease; known CNS metastases unless treated, are asymptomatic, are without evidence of radiological progression for at least 8 weeks, and have had no requirement for steroids or enzyme inducing anticonvulsants in the last 14 days prior to Screening.
* Abnormal pulmonary function within the previous 6 months, including pneumonitis, active pneumonitis, interstitial lung disease requiring the use of steroids, idiopathic pulmonary fibrosis, confirmed pleural effusion, severe dyspnea at rest or requiring supplementary oxygen therapy.
* Parenteral antibiotics within 14 days of the first dose of study drug.
* History of allogenic or solid organ transplant.
* Uncontrolled diabetes mellitus or other uncontrolled immune-related endocrinopathies in the opinion of the Investigator.
* Known human immunodeficiency virus (HIV) infection or active infection with hepatitis C.
* For known uncontrolled hepatitis B virus (HBV) infection:

  i. Anti-HBV therapy started before initiation of IMP and HBV viral load <2000 IU/mL (104 copies/mL) are eligible. The anti-HBV therapy should continue throughout the treatment period. ii. Positive anti-HBc, positive anti HBs, negative HBsAg, and HBV virus load without HBV therapy are eligible.
* Received a live-virus vaccination ≤14 days prior to first dose of study drug. Seasonal flu and other inactivated vaccines that do not contain live virus are permitted.
* Clinically significant bleeding within 2 weeks prior to initial THOR-707 dose (e.g., gastrointestinal bleeding, intracranial hemorrhage).
* Prior diagnosis of deep vein thrombosis or pulmonary embolism within 3 months.
* Severe or unstable cardiac condition within 6 months prior to starting study treatment, such as congestive heart failure (New York Heart Association Class III or IV), cardiac bypass surgery or coronary artery stent placement, angioplasty, cardiac ejection fraction below the lower limit of normal, unstable angina, medically uncontrolled hypertension (e.g. ≥160 mm Hg systolic or ≥100 mm Hg diastolic), uncontrolled cardiac arrhythmia requiring medication (≥ grade 2, according to NCI CTCAE v5.0), or myocardial infarction.
* History of non-pharmacologically induced prolonged corrected QT interval determined using Fridericia's formula (QTcF) > 450 milliseconds (msec) in males or > 470 msec in females.
* Known hypersensitivity or contraindications to any components of THOR-707, PEG, pegylated drugs, and E. coli derived-protein, checkpoint inhibitor, or anti-EGFR antibody for applicable cohorts.
* Active second malignancy, or history of previous malignancy that would impact the assessment of any study endpoints. Subjects with non-melanomatous skin cancer or cervical cancer that has been curatively surgically resected are eligible.
* Any serious medical condition (including pre-existing autoimmune disease or inflammatory disorder), laboratory abnormality, psychiatric condition, or any other significant or unstable concurrent medical illness that in the opinion of the Investigator would preclude protocol therapy or would make the subject inappropriate for the study.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through for at least 7 days (for Cohorts A, B, G, and H), at least 2 months (for Cohort D), or at least 4 months (for Cohorts C, E, and F) for females and for at least 3 days for males [corresponding to the time needed to eliminate study intervention] after the last dose of study intervention.
* Concurrent therapy with any other investigational agent, vaccine, or device. Concomitant participation in observational studies is acceptable after Sponsor approval.
* For Cohort D only: patients with symptomatic keratitis and/or symptomatic dry eye should be excluded from enrollment. Patients who wear contact lenses should be advised to avoid contact lenses use as it could result in keratitis.
* Subjects with baseline oxygen saturation <92% are not eligible for enrollment.
* For participants in Cohort H: Participants with uveal or ocular or desmoplastic metastatic melanoma.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Rate of Dose-Limiting Toxicities (DLTs)- Cohorts A, B, C, and D | Study Day 1 up to Day 29
  Based on toxicities observed
Maximum Tolerated Dose (MTD)- Cohorts A, B, C, and D | Study Day 1 up to Day 29
  Based on toxicities observed
Recommended Phase 2 Dose (RP2D)- Cohorts A, B, C, and D | Study Day 1 up to Day 29
  Based on toxicities observed
Number of participants with treatment emergent adverse events, serious adverse events, and laboratory abnormalities - Cohorts A, B, C, D, E, F, and G | Study Day 1 up to approximately 24 months
  Safety will be assessed by monitoring adverse events, clinical laboratory evaluations, vital signs, and ECG parameters.
Rate of Dose-Limiting Toxicities (DLTs) -Cohort G | Study Day 1 up to Day 42 (6 week-cycle)
  Based on toxicities observed
Recommended Phase 2 Dose (RP2D) of THOR-707- Cohort G | Study Day 1 up to Day 42 (6 week-cycle)
  Based on toxicities observed
Maximum Tolerated Dose (MTD)- Cohort G | Study Day 1 up to Day 42 (6 week-cycle)
  Based on toxicities observed
Objective Response Rate (ORR) according to RECIST version 1.1 -Cohort H | Study Day 1 up to approximately 24 months
  ORR, defined as the proportion of subjects with confirmed complete response (CR) or partial response (PR); a confirmed response is a response that persists on repeat-imaging ≥4 weeks after initial documentation of response.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) according to RECIST version 1.1 Cohort A, B, C, D, E, F, and G) | Study Day 1 up to approximately 24 months
  Defined as the proportion of subjects with confirmed complete response (CR) or partial response (PR); a confirmed response is a response that persists on repeat-imaging ≥4 weeks after initial documentation of response.
Duration of Response (DOR) according to RECIST version 1.1 | Study Day 1 up to approximately 24 months
  Defined as time from date of first objective response (either CR or PR) to first documentation of radiographic disease progression or death due to any cause, whichever occurs first.
Progression-Free Survival (PFS) according to RECIST version 1.1 | Study Day 1 until the date of first documented progression or date of death from any cause, assessed up to approximately 24 months
  Defined as the time from first dose of THOR-707 to first documentation of radiographic disease progression or death due to any cause, whichever occurs first.
Overall Survival according to RECIST version 1.1 | Study Day 1 up to time of death, assessed up to approximately 24 months
  Defined as the time from first dose of THOR-707 to the date of death due to any cause.
Time to Response (TTR) according to RECIST version 1.1 | Study Day 1 up to approximately 24 months
  Defined as the time from first dose of THOR-707 to first documentation of objective response (either CR or PR).
Disease Control Rate (DCR) according to RECIST version 1.1 | Study Day 1 up to approximately 24 months
  Defined as the proportion of subjects who have achieved confirmed CR, PR, or stable disease (SD) determined by Investigator per RECIST 1.1.
Clinical Benefit Rate (CBR) | Study Day 1 up to approximately 24 months
  Defined as the proportion of participants with clinical benefit i.e., confirmed CR or PR as BOR (is defined as the best overall response observed from the date of first IMP until disease progression, death, cut-off date or initiation of subsequent anti-cancer therapy, whichever occurs first), or SD lasting at least 6 months.
Number of participants with treatment emergent adverse events, serious adverse events, laboratory abnormalities -Cohort H | Study Day 1 up to approximately 24 months
  Safety will be assessed by monitoring adverse events, clinical laboratory evaluations, vital signs, and ECG parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (24):
- United States (7):
  - Investigational Site Number-1008, Scottsdale, Arizona
  - Investigational Site Number-1005, Denver, Colorado
  - Investigational Site Number-1004, Sarasota, Florida
  - Investigational Site Number-1003, Nashville, Tennessee
  - Investigational Site Number-1007, Dallas, Texas
  - Investigational Site Number-1002, Houston, Texas
  - Investigational Site Number-1001, San Antonio, Texas
- Investigational Site Number-7002, Buenos Aires, Argentina
- Australia (4):
  - Investigational Site Number-2004, New South Whales
  - Investigational Site Number-2001, Perth
  - Investigational Site Number-2002, Victoria
  - Investigational Site Number-2003, Victoria
- Chile (2):
  - Investigational Site Number- 6001, Santiago
  - Investigational Site Number-6002, Santiago
- Singapore (2):
  - Investigational Site Number-4002, Singapore
  - Investigational Site-4001, Singapore
- Spain (8):
  - Investigational Site Number-5001, Barcelona
  - Investigational Site Number-5006, Barcelona
  - Investigational Site Number-5007, Barcelona
  - Investigational Site Number-5002, Madrid
  - Investigational Site Number-5003, Madrid
  - Investigational Site Number-5004, Madrid
  - Investigational Site Number-5005, Madrid
  - Investigational Site Number-5105, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.

REFERENCES:
- See also: TCD16843 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25441&tenant=MT_SNY_9011